CLINICAL TRIAL: NCT06012591
Title: Implementation of WHO Standards for Improving the Quality of Maternal-neonatal Care
Brief Title: Implementation of WHO Standards for Improving Maternal and Newborn Care
Acronym: IMAgiNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC 16/22
Record Dates: First submitted 2023-03-28; First posted 2023-08-25 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-03

CONDITIONS: Perinatal Care
Keywords: maternal and newborn care; quality of care; quality improvement; WHO standards

STUDY DESIGN:
Intervention Model Description: Before-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WHO Standard implementation (Other)
  Interventions: Other: Quality improvement recommendations (action plans)

INTERVENTIONS:
Other: Quality improvement recommendations (action plans) — Developed and implemented at facility level to address key quality gaps emerging from the baseline assessment

SUMMARY:
High-quality respectful care around the time of childbirth is a fundamental aspect of human rights and, according to recent global estimates, could prevent more than 100,000 maternal deaths and 1.3 million neonatal deaths annually. Despite some maternal and newborn health indicators in high-income countries being better in comparison to low-income and middle-income countries, existing evidence shows that improvements are needed in the quality of care provided to women and newborns in every country.

In 2016, the World Health Organization (WHO) developed a framework and a list of Standards for improving the quality of maternal and newborn care (QMNC). The WHO Standards define a set of 318 Quality Measures, divided into three key domains - experience of care, provision of care and availability of resources - which can be used to assess the QMNC at facility level. The ongoing project, named IMAgiNE (Improving MAternal Newborn carE), includes all maternities hospitals of the FVG Region and aimed at improving the quality of maternal and neonatal health care in the region. Quality of care is assessed using two complementary perspectives (women and health workers), with two validated questionnaires including about 100 quality measures based on the WHO Standards. It provides data on both the baseline assessment and the Quality Improvement component (progresses made).

ELIGIBILITY:
Inclusion Criteria:

For women:

1. Women who give birth at the nine maternity hospitals of the Friuli Venezia Giulia (FVG) Region, Italy

For health workers

1. All health workers directly involved in maternal/neonatal care at facility level in the FVG Region (i.e. general physicians currently working in maternal or neonatal care, midwives, nurses, neonatologists, obstetrics and gynecology doctors, and medical residents )

Exclusion Criteria:

For women:

1. Age <18 years;
2. Stillbirth or neonatal death;
3. Psychiatric problems who may interfere with the telephone interview;
4. Hidden pregnancy or women whose child has been adopted or placed in foster care;
5. Refusal to participate.

For health workers

1. Refusal to participate;
2. Prolonged absence with unavailability during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 9000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Maternal and Newborn Care Index evaluated by women | At hospital discharge (assessed up to day 5)
  Evaluated by questionnaire
Quality of Maternal and Newborn Care Index evaluated by health professionals | At hospital discharge (assessed up to day 5)
  Evaluated by questionnaire

SECONDARY OUTCOMES:
Frequency of caesarean section | At hospital discharge (assessed up to day 5)
Frequency of episiotomy | At hospital discharge (assessed up to day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lazzerini, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (8):
- Italy (8):
  - Ospedale San Polo Monfalcone, Monfalcone, Gorizia
  - Ospedale di S. Antonio, San Daniele, Udine
  - Ospedale di San Vito al Tagliamento, San Vito al Tagliamento, Udine
  - Ospedale di S. Antonio Abate, Tolmezzo, Udine
  - Casa di Cura Policlinico San Giorgio, Pordenone
  - IRCCS Burlo Garofolo, Trieste
  - Ospedale di Palmanova, Udine
  - Presidio Ospedaliero Universitario Santa Maria della Misericordia, Udine